CLINICAL TRIAL: NCT03495687
Title: Peak Expiratory Flow and Thoracic Mobility in People With Fibromyalgia. A Cross Sectional Study.
Brief Title: Breathing and Chest Wall Mobility in People With Fibromyalgia.
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Sormland County Council, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: uppsala17
Record Dates: First submitted 2018-03-13; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Fibromyalgia
Keywords: Respiratory function; Spinal mobility; Chest expansion
MeSH Terms: conditions — Fibromyalgia; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine differences between respiratory function in female fibromyalgia patients and healthy controls. The study will also examine differences in spine mobility and pain intensity.

DETAILED DESCRIPTION:
Fibromyalgia is characterized by persistent widespread pain and affects approximately 1-3% of the general population. Fibromyalgia is a multifactorial syndrome and much research has been done and several interesting facts discovered. Still, the etiology is unknown. The autonomic nervous system may be the cause of several symptoms of this condition and a pattern of abnormal autonomous functions has been described . Besides the autonomous nerve system the respiratory system has also potential to impact various body organs mainly by altered blood gas chemistry. Deviant respiratory function in local pain condition as in cervical and lumbar spine has been reported. Respiratory function in generalized pain as in people with fibromyalgia has not been given much consideration.

This project is an observational cross sectional study with the purpose to examine respiratory function in a group of females with fibromyalgia and compare with age-matched controls. Peak expiratory flow (PEF), Chest mobility, spinal mobility and pain palpation where measured at the same visit. Data about smoking habits was registered and in patients also the duration of pain. Measurement of the subject's weight and height were recorded and the body mass index (BMI) was calculated. For evaluation of forced exhalation, a Wright peak expiratory flow meter was used. PEF was measured three times and the best result was recorded. Spinal mobility was measured by using the Cervico-thoracic ratio (CTR) method. The CTR measure was done in a sitting position with the subject instructed to sit in an upright posture and look straight in front of them. The spinous process of the seventh cervical vertebra (C7) was palpated as the referent point and a mark was made on the vertex followed by marks for each motion segment between C7 to the fifth thoracic vertebra (T5) by using a CTR measuring strip. Then the subjects were told to flex the chin and the trunk forward as much as possible. Again, the distance between C7 and T5 was measured and the difference between measurements in upright position and maximum flexed position was calculated in mm for each segment to a total sum for all segments from C7-T5. A tape measure was used to measure the mobility of the thorax at maximum inhalation and exhalation at the level of proc. Xiphoideus. Every measurement was performed three times and the best measurement was recorded. Manual palpation for pain was done over the upper thoracic spine in the same area as the spinal mobility was measured, with subjects lying prone on an examination table. A total of 20 locations were palpated from C7 to T5. First left side facets, and then left side costotransverse joints in the same segmental level. The same procedure was then used for the right side. Palpation was done with a force of approximately 4kg/sq cm (equating to blanching of the thumb or fingernail). After each point was palpated the subject estimated perceived pain on a visual analogue scale.

A ratio was also constructed by PEF (l / min) / chest expansion (cm) called expiratory-inspiratory ratio.

ELIGIBILITY:
Inclusion Criteria:

* Female diagnosed fibromyalgia according to American College of Rheumatology 1990 criteria
* Age 20-65 years
* Informed consent

Exclusion Criteria:

* trauma in neck-shoulder or thoracic region with prolonged symptoms during the last three month before examination
* severe illness (neurological e.g Parkinson disease, neuromuscular e.g Multiple sclerosis, respiratory e.g chronic obstructive pulmonary disease, muscle/skeletal disease e.g ankylosing spondylitis)
* Inability to understand or follow instructions
* Inability to participate at measurement sessions

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with diagnosed fibromyalgia and female healthy subjects included as controls.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow | Day 1
  maximum airflow achieved during expiration delivered with maximal force starting from the level of maximal lung inflation
Chest expansion | Day 1
  measures the thoracic circumference at the end of forced inspiration minus thoracic circumference at the end of forced expiration with a tape measure in the level of proc. xiphoideus.
Spinal mobility | Day 1
  Measure flexion mobility in the upper thoracic spine (C7-T5) by using the Cervico thoracic ratio method.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Peterson, MD PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No